CLINICAL TRIAL: NCT04914416
Title: OxxyneaGS: Single Blinded Randomized Study
Brief Title: Evaluation of OxxyneaGS in Acute Glycemic Regulation on Light Hyperglycemic Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fytexia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: OXXGS
Record Dates: First submitted 2021-05-28; First posted 2021-06-04 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Hyperglycemia, Postprandial
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Verum T1 (Placebo Comparator)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T2 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T3 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T4 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T5 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T6 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T7 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T8 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T9 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T10 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T11 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T12 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T13 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T14 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T15 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T16 (Experimental)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17
- Verum T17 (Placebo Comparator)
  Interventions: Dietary Supplement: Verum T1; Dietary Supplement: Verum T2; Dietary Supplement: Verum T3; Dietary Supplement: Verum T4; Dietary Supplement: Verum T5; Dietary Supplement: Verum T6; Dietary Supplement: Verum T7; Dietary Supplement: Verum T8; Dietary Supplement: Verum T9; Dietary Supplement: Verum T10; Dietary Supplement: Verum T11; Dietary Supplement: Verum T12; Dietary Supplement: Verum T13; Dietary Supplement: Verum T14; Dietary Supplement: Verum T15; Dietary Supplement: Verum T16; Dietary Supplement: Verum T17

INTERVENTIONS:
Dietary Supplement: Verum T1 — Verum T1 is a placebo: microcristalline cellulose. Daily dosage is 1000 mg in 3 capsules.
Dietary Supplement: Verum T2 — Verum T2 is a 11500AAIU/g white kidney bean extract. Daily dosage is 1000 mg in 3 capsules.
Dietary Supplement: Verum T3 — Verum T3 is a 11500AAIU/g white kidney bean extract. Daily dosage is 565 mg in 3 capsules
Dietary Supplement: Verum T4 — Verum T4 is a 17500AAIU/g white kidney bean extract. Daily dosage is 1000 mg in 3 capsules
Dietary Supplement: Verum T5 — Verum T5 is a 17500AAIU/g white kidney bean extract. Daily dosage is 371 mg in 3 capsules
Dietary Supplement: Verum T6 — Verum T6 is a 34200AAIU/g white kidney bean extract. Daily dosage is 1000 mg in 3 capsules
Dietary Supplement: Verum T7 — Verum T4 is a 34200AAIU/g white kidney bean extract. Daily dosage is 512 mg in 3 capsules
Dietary Supplement: Verum T8 — Verum T8 is a 34200AAIU/g white kidney bean extract. Daily dosage is 190 mg in 3 capsules.
Dietary Supplement: Verum T9 — Verum T9 is a polyphenol mix extract ( olive leaf, and blackcurrant extract). Daily dosage is 1000 mg in 3 capsules
Dietary Supplement: Verum T10 — Verum T10 is a polyphenol mix extract ( olive leaf, and blackcurrant extract). Daily dosage is 500 mg in 3 capsules
Dietary Supplement: Verum T11 — Verum T11 is a polyphenol mix extract ( olive leaf, pomelo, pomegranate, and blackcurrant extract). Daily dosage is 900 mg in 3 capsules
Dietary Supplement: Verum T12 — Verum T12 is a polyphenol mix extract ( olive leaf, pomelo, pomegranate, and blackcurrant extract). Daily dosage is 600 mg in 3 capsules
Dietary Supplement: Verum T13 — Verum T13 is a polyphenol mix extract ( olive leaf, pomelo, pomegranate, and/or blackcurrant extract) with white kidney bean extract. Daily dosage is 1000 mg in 3 capsules.
Dietary Supplement: Verum T14 — Verum T14 is a polyphenol mix extract ( olive leaf, pomelo, pomegranate, and/or blackcurrant extract) with white kidney bean extract. Daily dosage is 900 mg in 3 capsules.
Dietary Supplement: Verum T15 — Verum T15 is a polyphenol mix extract ( olive leaf, pomelo, pomegranate, and/or blackcurrant extract) with white kidney bean extract, Zinc, and, black currant leaf extracts. Daily dosage is 1000 mg in 3 capsules.
Dietary Supplement: Verum T16 — Verum T16 is a polyphenol mix extract ( olive leaf, pomelo, pomegranate, and/or blackcurrant extract) with white kidney bean extract, and Zinc. Daily dosage is 1000 mg in 3 capsules.
Dietary Supplement: Verum T17 — Verum T17 is a placebo: microcristalline cellulose. Daily dosage is 1000 mg in 3 capsules.

SUMMARY:
This study aims to evaluate and select the best combination of polyphenol and white kidney bean ingredients in the acute glycemic modulation after a complete meal by measuring blood glucose and insulin.

ELIGIBILITY:
Inclusion Criteria:

* Glycemia: 100-125mg/dL
* Both sexes
* Overweight BMI range (27-32)
* Age: 20-50 years old

Exclusion Criteria:

* Metabolic/Chronical disease
* Menopausal women
* Being pregnant, breastfeeding or wanting to have a baby
* Former obese with a history of yoyo effect
* Have been involved in a weight loss program in the past 12 months or subjected to weight reduction surgery
* Having started or quit smoking, having a high alcohol consumption
* Have in the past been in a long-term antibiotherapy (1 month or more) and/or a regular antibiotherapy in the past 12 months
* Allergy to olive, artichoke, black currant, grapefruit, grape, white kidney bean, olive, pomegranate.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Acute change in glycemia in response to a meal, by measuring glucose concentration in the blood at different time points | 8 hours

SECONDARY OUTCOMES:
Lipid profile evolution after a meal | 8 hours
Oxxidative stress variation after a meal, measured by oxidized/reduced glutathione (GSH/GSSG) | 8 hours
Acute change in insulinemia in response to a meal, by measuring insulin concentration in the blood at different time points | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Alcaraz Ramon, Principal Investigator — UCAM
Locations (1):
- UCAM, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No